CLINICAL TRIAL: NCT05565911
Title: The Relationship of Postoperative Morbidity / Mortality Rates of Patients With Pulmonary Hypertension With Risk Factors
Brief Title: Postoperative Morbidity / Mortality Rates of Patients With Pulmonary Hypertension
Acronym: PulmonaryHT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Begüm Nemika Gökdemir, Begüm Nemika Gökdemir, MD, Baskent University
Other Study IDs: 2022-03/1615
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: oPAP Should be > 25mmHg in Right Heart Catheterization at Rest; There Should be Patients Who Will Undergo Non-cardiac and Non-obstetric Surgery
Keywords: pulmonary hypertension; hemodinamic monitorization
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — this is an observational study, there is no intervention.

SUMMARY:
Pulmonary hypertension (PHT) is an oPAP ≥25 mmHg as assessed by right heart catheterization at rest. It is divided into 5 groups according to its etiology and mechanism. The first group is patients with pulmonary arterial hypertension due to various reasons (drugs, connective tissue diseases, etc.). Group 2 is classified as left heart failure, group 3 is due to chronic lung disease and hypoxemia, group 4 is due to pulmonary arterial obstruction (most commonly CTEPH), and group 5 is patients with pulmonary hypertension due to multifactorial unspecified causes.

In the pathophysiology, pulmonary hypertension occurs when the balance is disturbed by endothelial dysfunction, decrease in vasodilator mediators (NO, prostacyclin) and increase in vasoconstrictor mediators (endothelin-1, serotonin, thromboxan) in the vascular bed.

Perioperatively, patients with WHO functional classification >2, right ventricular hypertrophy, obese, chronic renal failure, previous PTE, COPD, diabetes mellitus are more prone to complications related to pulmonary hypertension. Although factors such as emergency surgery, intraoperative vasopressor use, delayed intubation, acidosis, and hyperthermia pave the way for postoperative pulmonary complications, attention should be paid to mortality and morbidity since they are also preventable factors.

Postoperatively, as a result of the supine position triggering bronchospasm with secretions, acute lung injury in addition to the existing comorbidity occurs. With the increase in respiratory workload, acute respiratory failure develops with symptoms such as hypoxemia and hypercarbia. Residual anesthesia, increased pain or prolonged mechanical ventilation time also decrease functional residual capacity, increasing the possibility of atelectasis development.

With the records we kept in our study, we aimed to show which complications the patients with pulmonary hypertension faced after their surgeries due to their underlying diseases and References ESC/ERC Guidelines Eurepean Heart Journal 2016; 37:67-119 Aguirre MA, et al. Advances in Anesthesia 2018;36: 201-30

DETAILED DESCRIPTION:
Our study will be carried out by recording the patients with PHT who underwent non-cardiac and non-obstetric surgeries at Başkent University Ankara Hospital between 11/10/2021 and 11/10/2023. It was planned to select the patients participating in our study on a voluntary basis and to include only the patients who agreed to participate in the study. Informed consent will be obtained by informing the patients before the application.

Both patient groups will be evaluated in the anesthesia polyclinic in the preoperative period. Routine blood tests will be done. It was planned as a cohort study. Depending on the surgery type of the patients, GA or RA will be applied as appropriate. The drugs in the standard anesthesia method will be administered to the patients. Standard monitoring and, if necessary, other invasive monitoring methods will be applied. Echocardiography evaluations, pulmonary function tests will be planned, and control evaluations will be requested at the 3rd, 6th and 1st postoperative months.

By the team in the postoperative recovery unit, hypoventilation (falling below breath per minute), apnea (episodes longer than 10 seconds), hypoxemia (SpO2<90, nasal O2 or Room Air), tachypnea, dyspnea, arrhythmia, chest pain, tachycardia, hypotension 30 minutes in terms of symptoms such as hypertension, laryngospasm, bronchospasm, subcostal retraction. They will be followed throughout. They will be evaluated in terms of analgesia control with Numeric Pain Score.

It will be evaluated in terms of postoperative pulmonary complications (tracheal reintubation) in the recovery unit and afterwards, extubation failure, pulmonary edema, and pneumothorax at the end of the case, and records will be kept.

ELIGIBILITY:
Inclusion Criteria:

* • Dinlenme halinde sağ kalp kateterizasyonu ile oPAB> 25mmHg olan hastalar,

  * Non-obstetrik ve non-kardiyak cerrahi geçirecek hastalar

Exclusion Criteria:

* • Dinlenme halinde sağ kalp kateterizasyonu ile oPAB< 25mmHg olan hastalar,

  * Obstetrik veya kardiyak cerrahi geçirecek hastalar

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Araştırma kapsamında pulmoner hipertansiyonu olan hastaların geçirecekleri cerrahilerde kendi hasta popülasyonlarına özel ne gibi risk faktörlerine sahip oldukları, tedavi olan ve olmayanlarda postoperatif komplikasyon gelişme sıklığının araştırılması planlanmaktadır
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of postoperative morbidity/mortality | 11/2021- 11/2023
  In this study, we investigated how the risk factors of patients with pulmonary hypertension can be evaluated and how the treatment plan can be arranged to prevent postoperative complications and reduce postoperative morbidity/mortality rates. We aim to compare the postoperative morbidity/mortality rates and complication frequency of patients who were evaluated and treated preoperatively with those who did not receive treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided